CLINICAL TRIAL: NCT00186563
Title: Proof-of-concept Study for Bio-marker Assay Validation in Humans
Brief Title: A Human In-vivo Model for the Detection of Inflammatory and Nociceptive Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin Angst (Other)
Responsible Party: Sponsor-Investigator, Martin Angst, Professor of Anesthesia, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 79723
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Skin Diseases
MeSH Terms: conditions — Skin Diseases

INTERVENTIONS:
Procedure: Micro-plasmapheresis

SUMMARY:
This study aims to establish a novel approach assisting the rational development of analgesic and anti-inflammatory drugs. In a first step we will test in healthy human volunteers whether proteins mediating inflammation and pain can be detected in an experimentally induced inflammatory skin lesion. Fluids that will be used to detect such proteins will be collected from the inflamed skin site via small porous catheters. We wish to establish the expression pattern of different proteins and correlate it with various tests assessing pain.

ELIGIBILITY:
Inclusion Criteria:1. Age between 21-60. 2. Skin type II or III according to the classification of Fitzpatrick (II: fair skin, always burns, sometimes tans, III: medium skin, sometimes burns, always tans).
 Exclusion Criteria:1. History of a significant systemic disease, a dermatological disease, bleeding disorder, or chronic pain.

2. Consumption of analgesic drugs. 3. Hypersensitivity to sunlight.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13

PRIMARY OUTCOMES:
Cytokine-release profile in response to inflammation, noxious heat, and asministration of a COX-inhibitor

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Angst, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States